CLINICAL TRIAL: NCT03441126
Title: Blood Culture Improvement Guidelines and Diagnostic Stewardship for Antibiotic Reduction in Critically Ill Children
Acronym: Bright STAR
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00147182
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Sepsis; Bacteremia
Keywords: Diagnostic Stewardship; Pediatric; Blood Culture Test
MeSH Terms: conditions — Sepsis; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multicenter Quality Improvement program: Locally developed and reliably implemented ICU Quality Improvement program to reduce blood culture use.
  Interventions: Other: Multicenter Quality Improvement program

INTERVENTIONS:
Other: Multicenter Quality Improvement program — Participating institutions will not participate in an intervention study. Sites will design and implement local QI programs to improve care within their unit. Local healthcare teams, who are interested in directly and immediately improving patient outcomes, will devise customized tools. The Bright STAR Team will assess the impact of these local QI initiatives on patient health outcomes, using data that are collected as part of the QI programs or through routine clinical care.

SUMMARY:
This study will test the hypothesis that reliable implementation of an evidence-based clinical practice guideline for evaluation of patients with signs and symptoms of sepsis will decrease antibiotic use in pediatric intensive care units (PICUs).

DETAILED DESCRIPTION:
The Bright STAR Collaborative (BSC), or Blood Culture Improvement Guidelines and Diagnostic Stewardship for Antibiotic Reduction in Critically Ill Children Collaborative, is a multicenter quality improvement program to reduce blood culture use within pediatric intensive care units. Investigators will use data collected by participating sites to determine whether reliable implementation of clinical practice guidelines for evaluation of patients with signs and symptoms of sepsis can decrease antibiotic use in pediatric intensive care units. Investigators will perform a quasi-experimental study to compare outcome data in pre- and post- periods.

Greater than or equal to 10 institutions will participate in this collaborative. Participating institutions will develop and implement an evidenced-based clinical decision-making tool as part of their quality improvement (QI) program in their pediatric intensive care unit (PICU).

Aim 1: To determine if reliable implementation of clinical practice guidelines for evaluation of patients with signs and symptoms of sepsis can decrease blood culture use in pediatric intensive care units.

Aim 2: To determine if reliable implementation of clinical practice guidelines for evaluation of patients with signs and symptoms of sepsis can decrease central line-associated bloodstream infections in pediatric intensive care units.

Aim 3. To determine if reliable implementation of clinical practice guidelines for evaluation of patients with signs and symptoms of sepsis can reduce antibiotic use and Clostridium difficile infection.

Aim 4. To determine whether a clinical practice guideline for evaluation of patients with signs and symptoms of sepsis in the PICU has an unintended consequence of patient harm.

Aim 5. To evaluate the implementation of a multi-institutional quality improvement initiative and identify strategies for successful scale-up and adoption of similar practice guidelines in other clinical settings.

Variables: blood cultures and central line-associated blood stream infections (CLABSIs), antibiotic use, , episodes of Clostridium difficile infection mortality, length of stay, ICU readmission, hospital readmission, episodes of sepsis, and episodes of septic shock.

Analyses: The analytic approach equates to estimating and comparing the blood culture incidence during the "baseline/pre-implementation" and "post-implementation" periods, using a generalized linear mixed model (GLMM) assuming a Poisson distribution for the monthly number of blood cultures with the monthly number of patient days as an offset. Similar analyses will be conducted to evaluate the incidence of blood cultures drawn from central lines and CLABSIs. Due to the expected low incidence of CLABSIs, investigators will define time in quarters, not months, for that outcome. Similar analyses will be performed for secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Institutions that plan to develop and implement a quality improvement program to reduce blood culture use in their ICUs

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICU patient populations from units that develop and implement a quality improvement program to reduce blood culture use
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Blood culture rate | Change in blood cultures per 100 patient days per month at 42 months
  The primary outcome of interest is blood culture rate in participating PICUs. A blood culture will be defined as any blood culture processed by the clinical microbiology laboratory.

SECONDARY OUTCOMES:
Central line-associated bloodstream infections (CLABSI). | 42 months
  The secondary outcome of interest is CLABSIs in participating PICUs. The outcome measurement will include a denominator of catheter days in the participating units.We will measure the change in CLABSI rate per month.
Broad spectrum antibiotic use | 42 months
  Use of broad spectrum antibiotics; Total antibiotic days per 1,000 patient days per quarter
Clostridium difficile infection | 42 months
  Incidence of infections per 1000 patient days per quarter
Mortality | 42 months
  Death per hospital total ICU admissions comparing pre and post-intervention periods
Length of ICU stay | 42 months
  Days in ICU; median number of days comparing pre and post-intervention periods
ICU readmission | 42 months
  Readmission to the ICU within 7 days of discharge. We will measure the change in rate of readmission per total ICU admissions comparing pre and post-intervention periods
Hospital readmission | 42 months
  Readmission to hospital within 7 days of discharge where we measured change in rate of hospital readmission comparing pre and post-intervention periods at
Sepsis | 42 months
  Defined by the following: International Classification of Diseases (ICD)-10 codes ; Admissions with ICD-10 coded sepsis per total ICU admissions
Septic shock | 42 months
  Defined by the following: ICD-10 codes; Admissions with ICD-10 coded septic shock per total ICU admissions

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Milstone, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - St. Louis Children's Hospital, Washington University, St Louis, Missouri
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - OHSU Doernbecher Children's Hospital, Portland, Oregon
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
We will not collect any. We will only gather summary-level non Patient Health Information (PHI) from participating sites.

REFERENCES:
- [Background] Woods-Hill CZ, Fackler J, Nelson McMillan K, Ascenzi J, Martinez DA, Toerper MF, Voskertchian A, Colantuoni E, Klaus SA, Levin S, Milstone AM. Association of a Clinical Practice Guideline With Blood Culture Use in Critically Ill Children. JAMA Pediatr. 2017 Feb 1;171(2):157-164. doi: 10.1001/jamapediatrics.2016.3153. PMID 27942705
- [Background] Xie A, Woods-Hill CZ, King AF, Enos-Graves H, Ascenzi J, Gurses AP, Klaus SA, Fackler JC, Milstone AM. Work System Assessment to Facilitate the Dissemination of a Quality Improvement Program for Optimizing Blood Culture Use: A Case Study Using a Human Factors Engineering Approach. J Pediatric Infect Dis Soc. 2019 Mar 28;8(1):39-45. doi: 10.1093/jpids/pix097. PMID 29165616
- [Derived] Woods-Hill CZ, Koontz DW, Xie A, Colantuoni EA, Sick-Samuels A, Miller MR, Arthur A, Aneja A, Kumar U, Milstone AM; Brigh T STAR authorship group. Diagnostic stewardship for blood cultures in the pediatric intensive care unit: lessons in implementation from the BrighT STAR Collaborative. Antimicrob Steward Healthc Epidemiol. 2024 Sep 25;4(1):e148. doi: 10.1017/ash.2024.416. eCollection 2024. PMID 39346668